CLINICAL TRIAL: NCT07065864
Title: Ketone Body Administration Impact on Work Capacity and Physiologic Reserve at Altitude
Brief Title: Ketone Esters for Optimization of Operator Performance in Hypoxia
Acronym: HVMN7
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida Institute for Human and Machine Cognition (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB-2021-0029; H9240519C0016 (Other: U.S. Special Operations Command)
Record Dates: First submitted 2025-06-10; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Hypoxia
Keywords: Hypoxia
MeSH Terms: conditions — Hypoxia | interventions — formic acid 4-(3-oxobutyl)phenyl ester

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of two interventions per visit: placebo and ketone
Who Masked: Participant
Masking Description: Participants are blinded to ketone or placebo consumption.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketone (Experimental): Ketone consumption prior to 24 minute submaximal bicycle ride at simulated 4500 meter altitude.
  Interventions: Dietary Supplement: Ketone ester
- Placebo (Placebo Comparator): steady state submaximal exercise (6 minutes each at 40, 50, and 60% of the peak power achieved at VO2max) at simulated 4500m after consuming the ketone ester or placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Ketone ester — Standardized light meal, questionnaires, blood measurements (finger stick), resting physiology and steady state submaximal exercise (6 minutes each at 40, 50, and 60% of the peak power achieved at VO2max) at simulated 4500m after consuming the ketone ester or placebo (in randomized order).
  Arms: Ketone
Other: Placebo — steady state submaximal exercise (6 minutes each at 40, 50, and 60% of the peak power achieved at VO2max) at simulated 4500m after consuming the ketone ester or placebo
  Arms: Placebo

SUMMARY:
The primary purpose of the study was to investigate effects of an orally administered ketone ester drink on endurance exercise performance during acute extreme hypoxia. Drinking this ketone supplement increases energy substrates known as ketone bodies in the blood, which may also act as metabolic signaling molecules. The ketone drink used in this study is recognized by the FDA as generally regarded as safe (GRAS). Some reports suggest that high ketone levels may enhance one's ability to tolerate hypoxia.

DETAILED DESCRIPTION:
High altitude environments limit oxygen availability in circulation and working tissues, leading to a decreased physiological reserve during physical exertion. Acute hypoxia elevates heart rate during submaximal work in a compensatory attempt, but decreases maximal heart rate progressively with increasing hypoxia. This contributes to a reduction in aerobic power (i.e. maximal rate of oxygen uptake, VO2max) an average of 6.3% per 1000m of elevation. Consumption of exogenous ketone bodies has been shown to enhance oxygen availability at rest at simulated altitudes up to 6100m, associated with better cognitive performance.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males 18 years of age or older (females are excluded because the 7th SFG consists only of males)
* Able to provide informed consent
* Able to perform the prescribed exercise and all study assessments
* Proficiency with the English language (reading, writing, speaking)

Exclusion Criteria:

* Any health or medical condition (e.g., cardiovascular, respiratory, musculoskeletal, neurologic) that would preclude exercise testing or potentially influence exercise performance, as determined by health and medical history questionnaire.
* Any condition that would preclude an accurate DXA body composition scan (e.g. joint replacement).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 17 (Actual)
Dates: Start 2023-08-04 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-11-14 (Actual)

PRIMARY OUTCOMES:
Evaluate submaximal exercise performance | 6.5 hours time commitment
  Evaluate submaximal exercise performance and physiologic reserve in hypoxia after consuming the ketone ester or placebo drink. Submaximal steady state VO2 relative to VO2max is the primary dependent variable.
  High altitude environments limit oxygen availability in circulation and working tissues, leading to a decreased physiological reserve during physical exertion. This contributes to a reduction in aerobic power (i.e. maximal rate of oxygen uptake, VO2max) an average of 6.3% per 1000m of elevation. Consumption of exogenous ketone bodies has been shown to enhance oxygen availability at rest at simulated altitudes up to 6100m, associated with better cognitive performance.

SECONDARY OUTCOMES:
Evaluate physiologic reserve in hypoxia | 6.5 hours time commitment
  Evaluate submaximal steady state heart rate (HR) exercise variables ( ↑HR that is affiliated with hypoxia).

CONTACTS AND LOCATIONS:
Locations (1):
- Florida Institute for Human and Machine Cognition, Pensacola, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
All data will be immediately de-identified and shared with participants.

DOCUMENTS (1):
  • Informed Consent Form (2023-04-18): https://cdn.clinicaltrials.gov/large-docs/64/NCT07065864/ICF_000.pdf